CLINICAL TRIAL: NCT04270305
Title: Study of Navigation Skills in Cerebral Palsy for Assessment and Rehabilitation in Immersive Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 308
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Walking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orientation (Experimental): Orientation training with GRAIL
  Interventions: Other: Orientation
- walking (Active Comparator): Walking training with GRAIL
  Interventions: Other: walking

INTERVENTIONS:
Other: Orientation — In the first group CP patients undergo a four week training with once daily sessions lasting 30 minutes. The treatment includes exercises to improve navigation competences and orientation. During walk in VR environment with labyrinths of increasing complexity. Exercises include abilities such as orienting in complex environments, perceiving distance and planning routes to distant locations. The presence of landmarks has been included in some exercises to facilitate allocentric orientation strategies.
  Arms: orientation
Other: walking — In the second group CP patients undergo a four week training with once daily sessions lasting 30 minutes. The treatment includes exercises to improve walking and balance abilities. Using engaging VR environments (e.g. transfer your load from the left to the right side to avoid obstacles while skiing; shoot balls at targets inside an area; walk in a forest as fast as possible; hit as many elves as possible by squatting, and so on). No exercises for orientation are included in this group.
  Arms: walking

SUMMARY:
Spatial navigation refers to the ability to maintain a sense of direction/location while moving around the environment so to find one's way. It includes abilities such as orienting in complex environments,perceiving distance and planning routes to distant locations as well as mentally representing the reciprocal relations of landmarks in space (Lawton, 2010; Wolbers & Hegarty 2010. Spatial navigation involves the precision in encoding multisensorial (visual, vestibular, proprioceptive)experiences, as well as to form mental representations to be used to guide behavior (Bianchini et al.,2014).

Cerebral Palsy (CP) is a neurodevelopmental disorder characterized by movement and posture disorders causing activity limitation. Impairment in many other functions is common in CP including visual spatial competences and spatial organization. In this study the investigators meant to explore the navigation and learning strategies in children with CP.

ELIGIBILITY:
Inclusion Criteria:.

* diagnosis of bilateral CP;
* age between 8 and 14 years old;
* severity of motor impairment classified in levels I, II and III, according to the Gross Motor Function Classification System (GMFCS) (Palisano et al., 1997)
* or according to the Manual Ability Classification System (MACS) (Eliasson et al., 2006);
* ability to follow instructions.

Exclusion Criteria:

* severe muscle spasticity and/or contracture,
* a diagnosis of severe learning disability,
* behavioral problems,
* visual or hearing difficulties that would affect the feasibility of proposed activities and/or compliance

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The Corsi Block Test | 1 month
  The Corsi Block Test (Orsini et al., 1987) assesses visuospatial memory and consists of a set of identical wooden blocks arranged more or less haphazardly on a desktop. The tester taps on a number of blocks in sequence, and the participant is asked to reproduce the tapped sequence, which is of variable length
The Labyrinth subtest of the WISC-III | 1 month
  The Labyrinth subtest of the WISC-III (Wechsler Intelligence Scale for Children, third version) consists of 10 paper-and-pencil tasks with increasing complexity (Weschler, 1991). The participant has to find the way out from the center of a 2-dimensional maze; it measures planning ability, perceptual organization, visualmotor coordination, and self-control

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No